CLINICAL TRIAL: NCT06527872
Title: The Evaluation Of Use of Belimumab in Routine Care SEttings in Lupus Nephritis (LN): the OBSErve-LN Study
Brief Title: Study to Assess Real-world Effectiveness of Belimumab for Treatment of Adults With LN
Acronym: OBSErve-LN
Status: Recruiting | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 216147
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Lupus Nephritis
Keywords: Belimumab; Lupus nephritis; OBSErve-LN; Renal function; Real world data
MeSH Terms: conditions — Lupus Nephritis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants cohort: Participants with active LN who initiated belimumab as per local label alongside standard therapy/ies under routine care conditions.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — Not Applicable since Observational Study
  Other Names: Observational Study

SUMMARY:
The purpose of the OBSErve-LN study is to assess the real-world use and effectiveness of belimumab in routine practice for the treatment of adults with active LN in multiple countries of interest. This study aims to provide the first long-term (up to 5 years) assessment of renal function preservation in belimumab treated participants.

DETAILED DESCRIPTION:
This is a Phase 4 study and will involve both prospective and retrospective data collection from participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants to provide a signed informed consent at the time of enrollment per protocol,
* Male or female aged 18 or over at initiation of belimumab,
* Participants received belimumab in any formulation (subcutaneous or intravenous) for the treatment of active LN prescribed as per local label in combination with standard immunosuppressive therapy/ies at initiation of belimumab,
* Participants initiated belimumab 6 to 24 months prior to study enrollment,
* Accessibility of medical records starting at belimumab initiation (including accessibility of medical records for the prior 12 months and confirmatory biopsy at any time prior to belimumab initiation),
* Biopsy-confirmed LN diagnosis at any time prior to belimumab initiation for treatment of LN
* Class III (focal LN) with or without Class V (membranous LN),
* Class IV (diffuse LN) with or without Class V,
* Class V.

Exclusion Criteria:

* Participants receiving renal replacement therapy (i.e., dialysis, kidney transplant, or those in end-stage kidney disease) at initiation of belimumab,
* Participant is concomitantly receiving another SLE targeted monoclonal antibody (MAb), or a MAb expected to compromise immune responses, at initiation of belimumab,
* Participants in a clinical trial during the observation period (with the exception of allowing participation in other non-interventional studies),
* Participant is pregnant at the initiation of belimumab,
* Participant with a kidney transplant at the initiation of belimumab,
* Participants will be excluded from the study if they are planning to become pregnant or are pregnant at study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include participants with lupus nephritis who initiated belimumab prescribed as per local label alongside standard therapy/ies under routine care conditions in the countries of interest.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2029-03-29 (Estimated); Study Completion 2029-03-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Maintaining Renal Function (Less than Equal to [<=] 30 Percentage [%] Decline in Estimated Glomerular Filtration Rate [eGFR] from the Initiation of Belimumab) and Not Requiring Renal Replacement Therapy | At Month 24
  Renal replacement therapy will involve participants requiring dialysis, kidney transplant, or those in end-stage kidney disease.

SECONDARY OUTCOMES:
Number of Participants Achieving Modified Partial Renal Response (<=20% Decline in eGFR and <=0.7 Urine Protein-Creatinine Ratio [uPCR]) and Modified Complete Renal Response (<=10% Decline in eGFR and <=0.5 uPCR) | At Months 24 and 60
Number of Participants Maintaining Renal Function (<=30% Decline in eGFR from the Initiation of Belimumab) and Not Requiring Renal Replacement Therapy (in Those that Remain Adherent to Belimumab) at Month 24 | At Month 24
  Renal replacement therapy will involve participants requiring dialysis, kidney transplant, or those in end-stage kidney disease.
Change in the Daily Dose of Steroid (in milligrams per day) from the Initiation of Belimumab | Baseline (Day 1) to Month 60
Estimated Glomerular Filtration Rate (eGFR) Slope over Time | Up to Month 60
Time to Achieving eGFR 30% and 40% Reduction | Up to Month 60
Time to Initiating Renal Replacement Therapy | Up to Month 60
  Renal replacement therapy will involve participants requiring dialysis, kidney transplant, or those in end-stage kidney disease.
Number of Participants Maintaining Renal Function (<=30% Decline in eGFR from the Initiation of Belimumab) and Not Requiring Renal Replacement Therapy | At Month 60
  Renal replacement therapy will involve participants requiring dialysis, kidney transplant, or those in end-stage kidney disease.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No